CLINICAL TRIAL: NCT03313037
Title: A PHASE 2, RANDOMIZED, DOUBLE-BLIND TRIAL TO EVALUATE THE SAFETY AND IMMUNOGENICITY OF A MULTIVALENT PNEUMOCOCCAL CONJUGATE VACCINE IN ADULTS 60 THROUGH 64 YEARS OF AGE
Brief Title: Trial to Evaluate the Safety and Immunogenicity of a Multivalent Pneumococcal Conjugate Vaccine in Adults 60 Through 64 Years of Age
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: B7471002
Record Dates: First submitted 2017-10-09; First posted 2017-10-18 (Actual); Results first posted 2019-12-26 (Actual); Last update posted 2019-12-26 (Actual); Status verified 2019-12

CONDITIONS: Pneumococcal Infections
MeSH Terms: conditions — Pneumococcal Infections | interventions — Vaccines, Combined; 13-valent pneumococcal vaccine; 23-valent pneumococcal capsular polysaccharide vaccine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Multivalent (Experimental): Pneumococcal conjugate vaccine
  Interventions: Biological: Multivalent; Other: Saline
- Control (Active Comparator): Prevnar 13 and PPSV23
  Interventions: Biological: Prevnar 13; Biological: PPSV23

INTERVENTIONS:
Biological: Multivalent — Pneumococcal conjugate vaccine
  Arms: Multivalent
Biological: Prevnar 13 — Pneumococcal conjugate vaccine
  Arms: Control
Biological: PPSV23 — Pneumococcal polysaccharide vaccine
  Other Names: Pneumovax 23
  Arms: Control
Other: Saline — Placebo
  Arms: Multivalent

SUMMARY:
This is a Phase 2, randomized, double-blinded study with a 2-arm parallel design. Healthy adults aged 60 through 64 years of age with no history of pneumococcal vaccination will be randomized equally to receive either a single intramuscular dose of multivalent pneumococcal conjugate vaccine followed 1 month later with a dose of saline or Prevnar 13 followed 1 month later with a dose of PPSV23 (control group).

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults >/= 60 to </=64 years of age (from the 60th birthday up to, but not including, the 65th birthday) at enrollment.
2. Healthy adults, including adults with preexisting stable disease, defined as disease not requiring significant change in therapy or requiring hospitalization within 3 months before receipt of investigational product, as determined by medical history, physical examination, laboratory screening, and clinical judgment of the investigator.
3. Female subjects who are not of childbearing potential.

Exclusion Criteria:

1. Previous vaccination with any licensed or investigational pneumococcal vaccine, or planned receipt through study participation.
2. History of microbiologically proven invasive disease caused by S pneumoniae.
3. Serious chronic disorder including metastatic malignancy, severe chronic obstructive pulmonary disease (COPD) requiring supplemental oxygen, end-stage renal disease with or without dialysis, clinically unstable cardiac disease, or any other disorder that, in the investigator's opinion, excludes the subject from participating in the study.

Ages: 60 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 444 (Actual)
Dates: Start 2017-10-10 (Actual); Primary Completion 2018-12-10 (Actual); Study Completion 2018-12-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (14):
- United States (14):
  - Anaheim Clinical Trials, LLC, Anaheim, California
  - Clinical Research of South Florida, Coral Gables, Florida
  - Avail Clinical Research, LLC, DeLand, Florida
  - Qps-Mra, Llc, South Miami, Florida
  - Clinical Research Atlanta, Stockbridge, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Heartland Research Associates, LLC, Wichita, Kansas
  - Lynn Health Science Institute, Oklahoma City, Oklahoma
  - Medical Research South, LLC, Charleston, South Carolina
  - Benchmark Research, Austin, Texas
  - Clinical Trials of Texas, Inc., San Antonio, Texas
  - Martin Diagnostic Clinic, Tomball, Texas
  - J. Lewis Research Inc. / Foothill Family Clinic Draper, Draper, Utah
  - J. Lewis Research, Inc. - Jordan River Family Medicine, South Jordan, Utah

IPD SHARING:
Plan to Share IPD: Yes
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.
URL: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- [Derived] Hurley D, Griffin C, Young M, Scott DA, Pride MW, Scully IL, Ginis J, Severs J, Jansen KU, Gruber WC, Watson W. Safety, Tolerability, and Immunogenicity of a 20-Valent Pneumococcal Conjugate Vaccine (PCV20) in Adults 60 to 64 Years of Age. Clin Infect Dis. 2021 Oct 5;73(7):e1489-e1497. doi: 10.1093/cid/ciaa1045. PMID 32716500
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7471002

RESULTS

PARTICIPANT FLOW:
Groups:
- 20vPnC Followed by Saline: Participants received a single 0.5 milliliter [mL] intramuscular injection of 20-valent pneumococcal conjugate vaccine (20vPnC) (Vaccination 1) on Day 1 followed by 0.5 mL of saline 1 month after Vaccination 1 (Vaccination 2). Participants were followed up to 12 months after Vaccination 1.
- 13vPnC Followed by PPSV23: Participants received a single 0.5 mL intramuscular injection of 13-valent pneumococcal conjugate vaccine (13vPnC) (Vaccination 1) on Day 1 followed by 0.5 mL of 23-valent pneumococcal polysaccharide vaccine (PPSV23) 1 month after Vaccination 1 (Vaccination 2). Participants were followed up to 12 months after Vaccination 1.
Period: Overall Study
Arm/Group | 20vPnC Followed by Saline | 13vPnC Followed by PPSV23
Started | 222 | 222
Safety Population | 221 | 222
Evaluable Immunogenicity Population(EIP) | 210 | 208
Completed | 202 | 202
Not Completed | 20 | 20
Not completed — Protocol Violation | 4 | 1
Not completed — Other | 1 | 1
Not completed — Withdrawal by Subject | 4 | 3
Not completed — No longer meets eligibility criteria | 1 | 7
Not completed — Lost to Follow-up | 9 | 8
Not completed — Randomized but not treated | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who had received 1 dose of 20vPnC or 13vPnC.
Groups:
- Total: Total of all reporting groups
Arm/Group | 20vPnC Followed by Saline | 13vPnC Followed by PPSV23 | Total
Number analyzed (Participants) | 221 | 222 | 443
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (1.40) | 62.0 (1.41) | 62.0 (1.41)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 115 | 133 | 248
  Male | 106 | 89 | 195
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 27 | 25 | 52
  Not Hispanic or Latino | 192 | 195 | 387
  Unknown or Not Reported | 2 | 2 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 2 | 3
  Asian | 8 | 7 | 15
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 1
  Black or African American | 37 | 46 | 83
  White | 169 | 165 | 334
  More than one race | 4 | 2 | 6
  Unknown or Not Reported | 1 | 0 | 1

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Local Reactions Within 10 Days After Vaccination 1
Description: Local reactions included pain at injection site, swelling and redness recorded by participants in an electronic diary (e-diary). Redness and swelling were measured and recorded in measuring device units. 1 measuring device unit=0.5 centimeter (cm). Redness and swelling were graded as mild: greater than (>) 2.0 to 5.0 centimeter (cm), moderate: 5.5 to 10.0 cm and severe: greater than or equal to (>=) 10.5 cm. Pain was graded as mild: did not interfere with activity, moderate: interfered with activity and severe: prevented daily activity.
Time Frame: within 10 days after Vaccination 1
Population: Safety analysis set included all participants who had received 1 dose of 20vPnC or 13vPnC. Here "Overall number of participants analyzed" signifies participants who were evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 20vPnC Followed by Saline | 13vPnC Followed by PPSV23
Number analyzed (Participants) | 220 | 222
percentage of participants
  Redness: Mild | 7.3 [4.2 to 11.5] | 3.6 [1.6 to 7.0]
  Redness: Moderate | 3.6 [1.6 to 7.0] | 3.2 [1.3 to 6.4]
  Redness: Severe | 0.5 [0.0 to 2.5] | 0 [0.0 to 1.6]
  Swelling: Mild | 7.7 [4.6 to 12.1] | 7.7 [4.5 to 12.0]
  Swelling: Moderate | 5.5 [2.8 to 9.3] | 3.6 [1.6 to 7.0]
  Swelling: Severe | 0 [0.0 to 1.7] | 0 [0.0 to 1.6]
  Pain at injection site: Mild | 46.8 [40.1 to 53.6] | 43.7 [37.1 to 50.5]
  Pain at injection site: Moderate | 10.9 [7.1 to 15.8] | 9.5 [6.0 to 14.1]
  Pain at injection site: Severe | 0 [0.0 to 1.7] | 0.5 [0.0 to 2.5]

2. Primary Outcome: Percentage of Participants With Systemic Events Within 7 Days After Vaccination 1
Description: Systemic events included fever, fatigue, headache, muscle pain and joint pain, recorded by participants in an e-diary. Fever was categorized as: >=38.0 degrees Celsius (C), >=38.0 to 38.4 degrees C, >38.4 to 38.9 degrees C, >38.9 to 40.0 degrees C and >40.0 degrees C. Fatigue, headache, muscle pain and joint pain were graded as mild: no interference with activity, moderate: some interference with activity and severe: prevents daily routine activity.
Time Frame: within 7 days after Vaccination 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 20vPnC Followed by Saline | 13vPnC Followed by PPSV23
Number analyzed (Participants) | 220 | 222
percentage of participants
  Fever: >=38.0 degree C | 0 [0.0 to 1.7] | 0.5 [0.0 to 2.5]
  Fever: >=38.0 to 38.4 degree C | 0 [0.0 to 1.7] | 0.5 [0.0 to 2.5]
  Fever: >38.4 to 38.9 degree C | 0 [0.0 to 1.7] | 0 [0.0 to 1.6]
  Fever: >38.9 to 40.0 degree C | 0 [0.0 to 1.7] | 0 [0.0 to 1.6]
  Fever: >40.0 degree C | 0 [0.0 to 1.7] | 0 [0.0 to 1.6]
  Fatigue: Mild | 19.1 [14.1 to 24.9] | 18.0 [13.2 to 23.7]
  Fatigue: Moderate | 11.4 [7.5 to 16.3] | 10.4 [6.7 to 15.1]
  Fatigue: Severe | 0.5 [0.0 to 2.5] | 1.8 [0.5 to 4.5]
  Headache: Mild | 16.8 [12.1 to 22.4] | 18.0 [13.2 to 23.7]
  Headache: Moderate | 3.6 [1.6 to 7.0] | 5.4 [2.8 to 9.3]
  Headache: Severe | 0.5 [0.0 to 2.5] | 0.9 [0.1 to 3.2]
  Muscle pain: Mild | 32.7 [26.6 to 39.4] | 27.0 [21.3 to 33.4]
  Muscle pain: Moderate | 10.5 [6.7 to 15.3] | 9.5 [6.0 to 14.1]
  Muscle pain: Severe | 0 [0.0 to 1.7] | 0 [0.0 to 1.6]
  Joint pain: Mild | 9.5 [6.0 to 14.2] | 8.1 [4.9 to 12.5]
  Joint pain: Moderate | 5.5 [2.8 to 9.3] | 5.9 [3.2 to 9.8]
  Joint pain: Severe | 0 [0.0 to 1.7] | 0.5 [0.0 to 2.5]

3. Primary Outcome: Percentage of Participants With Adverse Events (AEs) Within 1 Month After Vaccination 1
Description: An AE was any untoward medical occurrence in a participant who received investigational product without regard to possibility of causal relationship. AEs included both serious and non-serious adverse events. Serious adverse event (SAE) was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: within 1 month after Vaccination 1 (up to 35 days)
Population: Safety analysis set included all participants who had received 1 dose of 20vPnC or 13vPnC.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 20vPnC Followed by Saline | 13vPnC Followed by PPSV23
Number analyzed (Participants) | 221 | 222
percentage of participants | 12.2 [8.2 to 17.3] | 13.1 [8.9 to 18.2]

4. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) or Newly Diagnosed Chronic Medical Conditions (NDCMCs) Within 6 Months After Vaccination 1
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. SAE was an AE resulting in any of the following outcomes or deemed significant for any other reason: death; initial or prolonged inpatient hospitalization; life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly. An NDCMC was defined as a disease or medical condition, not previously identified, that is expected to be persistent or is otherwise long-lasting in its effects. Percentage of participants with either SAE or NDCMCs during the specified duration are reported.
Time Frame: within 6 months after Vaccination 1 (up to 196 days)
Population: Safety analysis set included all participants who had received 1 dose of 20vPnC or 13vPnC.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 20vPnC Followed by Saline | 13vPnC Followed by PPSV23
Number analyzed (Participants) | 221 | 222
percentage of participants | 5.4 [2.8 to 9.3] | 4.5 [2.2 to 8.1]

5. Primary Outcome: Percentage of Participants With Serious Adverse Events (SAEs) or Newly Diagnosed Chronic Medical Conditions (NDCMCs) Within 12 Months After Vaccination 1
Description: as for outcome 4
Time Frame: within 12 months after Vaccination 1 (up to 378 days)
Population: Safety analysis set included all participants who had received 1 dose of 20vPnC or 13vPnC.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | 20vPnC Followed by Saline | 13vPnC Followed by PPSV23
Number analyzed (Participants) | 221 | 222
percentage of participants | 10.0 [6.3 to 14.7] | 6.3 [3.5 to 10.4]

6. Secondary Outcome: Serotype-Specific Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Titres (GMTs) 1 Month After Vaccination 1: 13 Common Serotypes in 13vPnC
Description: Antibody-mediated serum OPA against the 13 common pneumococcal serotypes specific to 13vPnC (serotypes 1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F and 23F) were measured using a pneumococcal OPA assay. Results were expressed as OPA GMTs. Assay results below the lower limit of quantitation (LLOQ) were set to 0.5*LLOQ in the analysis.
Time Frame: 1 month after Vaccination 1
Population: EIP: participants with no major protocol deviations, received assigned vaccine, blood drawn within 27 to 49 days after Vaccination 1 or 2, had OPA titres for at least 1 serotype either 1 month after Vaccination 1 or 2. 'Number analyzed' = Participants evaluable for this outcome measure at specified rows.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer (1/dilution)
Arm/Group | 20vPnC Followed by Saline | 13vPnC Followed by PPSV23
Number analyzed (Participants) | 210 | 208
Titer (1/dilution)
  Serotype 1: number analyzed (Participants) | 205 | 205
  Serotype 1 | 302 [239.6 to 381.4] | 454 [352.6 to 584.5]
  Serotype 3: number analyzed (Participants) | 208 | 204
  Serotype 3 | 51 [43.2 to 61.2] | 64 [54.1 to 76.7]
  Serotype 4: number analyzed (Participants) | 202 | 200
  Serotype 4 | 876 [676.8 to 1134.7] | 1153 [883.3 to 1504.1]
  Serotype 5: number analyzed (Participants) | 204 | 202
  Serotype 5 | 144 [113.3 to 183.2] | 215 [168.7 to 274.4]
  Serotype 6A: number analyzed (Participants) | 205 | 199
  Serotype 6A | 1907 [1492.7 to 2436.2] | 2440 [1848.9 to 3219.9]
  Serotype 6B: number analyzed (Participants) | 201 | 202
  Serotype 6B | 2006 [1591.4 to 2527.5] | 2218 [1716.9 to 2865.1]
  Serotype 7F: number analyzed (Participants) | 207 | 204
  Serotype 7F | 1581 [1361.6 to 1836.0] | 1936 [1651.1 to 2269.6]
  Serotype 9V: number analyzed (Participants) | 207 | 203
  Serotype 9V | 1164 [949.6 to 1428.0] | 1612 [1311.4 to 1981.4]
  Serotype 14: number analyzed (Participants) | 206 | 204
  Serotype 14 | 1114 [905.0 to 1371.4] | 1282 [1017.4 to 1614.9]
  Serotype 18C: number analyzed (Participants) | 204 | 203
  Serotype 18C | 1322 [1053.2 to 1658.9] | 1660 [1335.1 to 2064.5]
  Serotype 19A: number analyzed (Participants) | 207 | 203
  Serotype 19A | 943 [783.5 to 1136.1] | 1137 [936.5 to 1379.4]
  Serotype 19F: number analyzed (Participants) | 204 | 205
  Serotype 19F | 455 [349.2 to 592.2] | 738 [582.1 to 936.5]
  Serotype 23F: number analyzed (Participants) | 206 | 205
  Serotype 23F | 408 [293.0 to 568.0] | 509 [377.3 to 687.1]

7. Secondary Outcome: Serotype-Specific Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Titres (GMTs) 1 Month After Any Vaccination: 7 Additional Serotypes in 20vPnC
Description: Antibody-mediated serum OPA against the 7 additional pneumococcal serotypes (8, 10A, 11A, 12F, 15B, 22F, 33F) were measured using a pneumococcal OPA assay. Results were expressed as OPA GMTs. Assay results below the LLOQ were set to 0.5*LLOQ in the analysis.
Time Frame: 1 month after Vaccination 1 for 20vPnC followed by saline reporting group; 1 month after Vaccination 2 for 13vPnC followed by PPSV23 reporting group
Population: as for outcome 6
Measure: Geometric Mean (95% Confidence Interval); unit: Titer (1/dilution)
Arm/Group | 20vPnC Followed by Saline | 13vPnC Followed by PPSV23
Number analyzed (Participants) | 210 | 208
Titer (1/dilution)
  Serotype 8: number analyzed (Participants) | 207 | 200
  Serotype 8 | 740 [598.0 to 915.7] | 1150 [944.4 to 1401.6]
  Serotype 10A: number analyzed (Participants) | 201 | 197
  Serotype 10A | 2604 [2096.4 to 3234.4] | 988 [731.2 to 1335.5]
  Serotype 11A: number analyzed (Participants) | 197 | 200
  Serotype 11A | 3210 [2613.2 to 3943.8] | 3007 [2443.0 to 3700.3]
  Serotype 12F: number analyzed (Participants) | 200 | 191
  Serotype 12F | 6571 [5022.2 to 8597.3] | 4290 [3190.8 to 5769.1]
  Serotype 15B: number analyzed (Participants) | 205 | 200
  Serotype 15B | 1889 [1434.7 to 2488.3] | 720 [530.8 to 975.9]
  Serotype 22F: number analyzed (Participants) | 201 | 189
  Serotype 22F | 6286 [5025.0 to 7863.2] | 3513 [2824.8 to 4367.7]
  Serotype 33F: number analyzed (Participants) | 185 | 181
  Serotype 33F | 5584 [4374.1 to 7128.0] | 3940 [3136.2 to 4950.9]

8. Secondary Outcome: Serotype-specific Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Fold Rise (GMFR) From Pre-Vaccination 1 to 1 Month Post-Vaccination 1: 13 Common Serotypes in 13vPnC
Description: GMFR for the 13 pneumococcal serotypes (1, 3, 4, 5, 6A, 6B, 7F, 9V, 14, 18C, 19A, 19F, and 23F) from before Vaccination 1 to one month after Vaccination 1 were calculated as the mean of the difference of logarithmically transformed OPA results (after vaccination - before vaccination) and transform back to the original scale. GMFRs were calculated using data from participants with non-missing OPA results at both time points. Assay results below the LLOQ were set to 0.5*LLOQ in the analysis.
Time Frame: before Vaccination 1 to one month after Vaccination 1
Population: EIP: participants with no major protocol deviations, received assigned vaccine, blood drawn within 27 to 49 days after Vaccination 1 or 2, had OPA titres for at least 1 serotype either 1 month after Vaccination 1 or 2. 'Number analyzed' = Number of participants with non-missing OPA results at both time points at specified rows.
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | 20vPnC Followed by Saline | 13vPnC Followed by PPSV23
Number analyzed (Participants) | 210 | 208
fold rise
  Serotype 1: number analyzed (Participants) | 204 | 205
  Serotype 1 | 21.2 [16.96 to 26.60] | 33.5 [25.77 to 43.65]
  Serotype 3: number analyzed (Participants) | 208 | 204
  Serotype 3 | 6.0 [5.02 to 7.23] | 7.1 [5.85 to 8.60]
  Serotype 4: number analyzed (Participants) | 195 | 193
  Serotype 4 | 37.8 [27.40 to 52.10] | 51.0 [36.04 to 72.27]
  Serotype 5: number analyzed (Participants) | 204 | 202
  Serotype 5 | 8.3 [6.55 to 10.54] | 11.6 [9.09 to 14.86]
  Serotype 6A: number analyzed (Participants) | 196 | 191
  Serotype 6A | 58.6 [44.15 to 77.73] | 68.6 [49.49 to 95.20]
  Serotype 6B: number analyzed (Participants) | 193 | 188
  Serotype 6B | 29.6 [22.56 to 38.96] | 38.8 [28.52 to 52.66]
  Serotype 7F: number analyzed (Participants) | 195 | 194
  Serotype 7F | 12.2 [9.86 to 15.22] | 15.8 [12.57 to 19.82]
  Serotype 9V: number analyzed (Participants) | 202 | 196
  Serotype 9V | 7.7 [6.15 to 9.57] | 10.1 [7.95 to 12.74]
  Serotype 14: number analyzed (Participants) | 198 | 198
  Serotype 14 | 8.5 [6.35 to 11.26] | 9.6 [7.20 to 12.89]
  Serotype 18C: number analyzed (Participants) | 200 | 195
  Serotype 18C | 26.8 [19.96 to 35.85] | 35.2 [26.02 to 47.50]
  Serotype 19A: number analyzed (Participants) | 204 | 202
  Serotype 19A | 23.3 [17.96 to 30.19] | 30.9 [23.70 to 40.37]
  Serotype 19F: number analyzed (Participants) | 201 | 204
  Serotype 19F | 11.8 [8.93 to 15.47] | 18.4 [14.19 to 23.87]
  Serotype 23F: number analyzed (Participants) | 205 | 203
  Serotype 23F | 33.6 [24.19 to 46.54] | 39.8 [28.85 to 54.88]

9. Secondary Outcome: Serotype-specific Pneumococcal Opsonophagocytic Activity (OPA) Geometric Mean Fold Rise (GMFR) From Pre-Vaccination 1 to 1 Month Post Any Vaccination: 7 Additional Serotypes in 20vPnC
Description: GMFR for 7 additional pneumococcal serotypes (8, 10A, 11A, 12F, 15B, 22F, 33F) from before Vaccination 1 to one month after either Vaccination 1 (20vPnC) or Vaccination 2 (PPSV23) were calculated as the mean of the difference of logarithmically transformed OPA results (after vaccination - before vaccination) and transform back to the original scale. GMFRs were calculated using data from participants with non-missing OPA results at both time points. Assay results below the LLOQ were set to 0.5*LLOQ in the analysis.
Time Frame: before Vaccination 1 to 1 month after Vaccination 1 for 20vPnC followed by saline reporting group; before Vaccination 1 to 1 month after Vaccination 2 for 13vPnC followed by PPSV23 reporting group
Population: EIP: participants with no protocol deviations, received assigned vaccine, blood drawn within 27 to 49 days after Vaccination 1 or 2, had OPA titres for at least 1 serotype either 1 month after Vaccination 1 or 2. 'Number analyzed' = Number of Participants with non-missing OPA results at both time points at specified row.
Measure: Geometric Mean (95% Confidence Interval); unit: fold rise
Arm/Group | 20vPnC Followed by Saline | 13vPnC Followed by PPSV23
Number analyzed (Participants) | 210 | 208
fold rise
  Serotype 8: number analyzed (Participants) | 203 | 196
  Serotype 8 | 37.1 [27.71 to 49.71] | 56.9 [42.90 to 75.46]
  Serotype 10A: number analyzed (Participants) | 192 | 188
  Serotype 10A | 49.3 [35.18 to 68.95] | 17.1 [12.15 to 24.15]
  Serotype 11A: number analyzed (Participants) | 190 | 175
  Serotype 11A | 11.2 [8.16 to 15.31] | 9.8 [7.41 to 13.06]
  Serotype 12F: number analyzed (Participants) | 183 | 183
  Serotype 12F | 113.4 [81.47 to 157.90] | 77.0 [55.04 to 107.64]
  Serotype 15B: number analyzed (Participants) | 201 | 195
  Serotype 15B | 57.1 [41.74 to 78.07] | 21.3 [15.30 to 29.71]
  Serotype 22F: number analyzed (Participants) | 184 | 178
  Serotype 22F | 55.4 [38.88 to 79.01] | 20.3 [14.69 to 27.96]
  Serotype 33F: number analyzed (Participants) | 168 | 169
  Serotype 33F | 14.0 [9.96 to 19.62] | 8.9 [6.67 to 11.84]

ADVERSE EVENTS:
Time Frame: Local reactions: within 10 days after vaccination (systematic assessment), Systemic events: within 7 days after vaccination (systematic assessment), Non serious AEs: Baseline up to 1 month after Vaccination 1 (up to 35 days), SAEs: Baseline up to 12 months after Vaccination 1 (up to 378 days)
Description: Same event may appear as both an adverse event (AE) and serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in 1 participant and as non-serious in another, or a participant may have experienced both a serious and non-serious event. Safety population was analyzed.
Arm/Group | 20vPnC Followed by Saline | 13vPnC Followed by PPSV23
All-Cause Mortality (participants affected / at risk) | 0/221 | 0/222
Serious Adverse Events (participants affected / at risk) | 9/221 | 11/222
Other Adverse Events (participants affected / at risk) | 162/221 | 164/222
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 20vPnC Followed by Saline (N=221) | 13vPnC Followed by PPSV23 (N=222)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Cardiomyopathy (Cardiac disorders) | 0 | 1
Chest pain (General disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1
Cellulitis staphylococcal (Infections and infestations) | 1 | 0
Meningitis pneumococcal (Infections and infestations) | 0 | 1
Septic shock (Infections and infestations) | 1 | 0
Head injury (Injury, poisoning and procedural complications) | 0 | 1
Lower limb fracture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Spindle cell sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Uterine cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 2
Lacunar infarction (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 1 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 20vPnC Followed by Saline (N=221) | 13vPnC Followed by PPSV23 (N=222)
Injection site pruritus (General disorders) | 0 | 1
Acute sinusitis (Infections and infestations) | 1 | 2
Bronchitis (Infections and infestations) | 2 | 0
Gastroenteritis (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 3 | 0
Tooth infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 7 | 5
Fall (Injury, poisoning and procedural complications) | 0 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Dizziness (Nervous system disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Lymphadenopathy (Blood and lymphatic system disorders) | 1 | 0
Deafness unilateral (Ear and labyrinth disorders) | 0 | 1
Hypothyroidism (Endocrine disorders) | 1 | 0
Dental caries (Gastrointestinal disorders) | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 0
Chest pain (General disorders) | 0 | 1
Fatigue (General disorders) | 68 | 67
Injection site hypersensitivity (General disorders) | 1 | 0
Injection site pain (General disorders) | 1 | 1
Injection site pain (General disorders) | 127 | 119
Pyrexia (General disorders) | 0 | 1
Swelling (General disorders) | 29 | 25
Gastroenteritis viral (Infections and infestations) | 1 | 1
Gingivitis (Infections and infestations) | 0 | 1
Laryngitis viral (Infections and infestations) | 0 | 1
Nasopharyngitis (Infections and infestations) | 0 | 2
Urinary tract infection (Infections and infestations) | 2 | 0
Vaginal infection (Infections and infestations) | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 0 | 1
Muscle strain (Injury, poisoning and procedural complications) | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 0 | 2
Gout (Metabolism and nutrition disorders) | 1 | 0
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 33 | 32
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 95 | 81
Headache (Nervous system disorders) | 1 | 0
Headache (Nervous system disorders) | 46 | 54
Lumbar radiculopathy (Nervous system disorders) | 1 | 0
Presyncope (Nervous system disorders) | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0
Asthma (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Sinus congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Upper respiratory tract congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Erythema (General disorders) | 25 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2017-07-20): https://cdn.clinicaltrials.gov/large-docs/37/NCT03313037/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-31): https://cdn.clinicaltrials.gov/large-docs/37/NCT03313037/SAP_001.pdf